CLINICAL TRIAL: NCT02192255
Title: An Intervention to Feedback 'Early' Non-Adherence Data to ImproveCardiovascular Disease Risk Factor Outcomes in Patients With Diabetes
Brief Title: SUPREME-DM (Diabetes Mellitis) Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-018
Record Dates: First submitted 2014-06-12; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes
Keywords: diabetes type 2; primary care; chronic disease care improvement; adherence, randomized trial; BP control; lipid control; glucose control; natural language processing.
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention phone call (Experimental): The intervention arm consisted of one protocol-structured telephone call from an interventionist who was a nurse health manager (1 site), diabetes educator or diabetes educator trainee (1 site), or pharmacist (2 sites). Interventionists followed the same structured telephone interview protocol to ascertain whether the subject had started taking the new prescription. Those taking the new medication as prescribed received positive reinforcement. Those who either had not filled the prescription or were not taking the medication as directed, were asked about reasons for nonadherence and assisted in identifying and resolving barriers. The median call lasted < than 5 minutes, and up to 3 call attempts were made. Most intervention calls occurred within 2 to 6 weeks after the prescription date.
  Interventions: Behavioral: Intervention Phone Call
- Control arm - usual care (No Intervention): Those in the control arm received usual care.

INTERVENTIONS:
Behavioral: Intervention Phone Call — The intervention arm consisted of one protocol-structured telephone call from an interventionist who was a nurse health manager (1 site), diabetes educator or diabetes educator trainee (1 site), or pharmacist (2 sites). Interventionists followed the same structured telephone interview protocol to ascertain whether the subject had started taking the new prescription. Those taking the new medication as prescribed received positive reinforcement. Those who either had not filled the prescription or were not taking the medication as directed, were asked about reasons for nonadherence and assisted in identifying and resolving barriers. The median call lasted < than 5 minutes, and up to 3 call attempts were made. Most intervention calls occurred within 2 to 6 weeks after the prescription date.
  Arms: Intervention phone call

SUMMARY:
This multisite pragmatic clinical trial was designed to assess the effectiveness of a single scripted telephone call to diabetes patients who (a) were currently above recommended clinical goals for glucose, blood pressure, or lipids, and (b) had recently been prescribed a new medication for that specific clinical domain. The goals of the intervention were to improve primary adherence and persistence to the newly prescribed medication and to improve control of glucose, blood pressure, and lipids.

DETAILED DESCRIPTION:
This randomized trial tested the hypothesis that a telephone contact with a patient recently prescribed a new medication for uncontrolled glycated hemoglobin (A1c), blood pressure, or low-density lipoprotein cholesterol would improve (a) primary medication adherence, (b) medication persistence, (c) medication possession ratio, and (d) A1c, blood pressure or low-density lipoprotein cholesterol control. This study was part of the larger Agency for Healthcare Research and Quality funded SUPREME-DM study. The clinical trial reported here was coordinated and led by HealthPartners Institute for Education and Research, while data collection was coordinated through Kaiser Permanente Northwest and analysis was conducted at Kaiser Permanente Colorado. The clinical intervention sites for this study included Kaiser Permanente Northern California, Group Health Cooperative, Marshfield Clinic, and Geisinger Clinic.

ELIGIBILITY:
Inclusion Criteria:

* At each clinical intervention site, study subjects were selected if they:

  * were age 18-75 years
  * met study criteria for diabetes mellitus before study enrollment
  * received clinical care at a designated clinic or medical center involved in this study for at least 15 months before enrollment
  * were prescribed a new class of medication (not filled in the past 180 days) for A1c, BP, or LDL that was uncontrolled at the time of medication prescription (A1c>=8%, systolic BP>= 140 mm Hg, or LDL >=100 mg/dL).

Exclusion Criteria:

* Study subjects were excluded if they were younger than 18 years of age
* Older than 75 years of age
* Did not have evidence of diabetes mellitus prior to study enrollment
* Were not receiving care at a clinic site involved in this study for at least 15 months before enrollment
* Did not have prescribed a new class of medication for uncontrolled A1c, BP or LDL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2378 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
60 day Medication Adherence | 60 days
  In a pragmatic randomized trial, we randomly assigned 2,378 adults with diabetes mellitus who were recently prescribed a new class of medication for elevated glycated hemoglobin (A1c) >= 8%, blood pressure >= 140/90 mm Hg, or low-density lipoprotein cholesterol >=100 mg/dL, to receive (a) one scripted telephone call from a diabetes educator or clinical pharmacist to identify and address nonadherence to the new medication or (b) usual care. Hierarchical linear and logistic regression models were used to assess impact on (a) first medication fill within 60 days of prescription,
120 day medication adherence | 120 days
  In a pragmatic randomized trial, we randomly assigned 2,378 adults with diabetes mellitus who were recently prescribed a new class of medication for elevated glycated hemoglobin (A1c) >= 8%, Blood pressure >= 140/90 mm Hg, or low-density lipoprotein cholesterol >=100 mg/dL, to receive (a) one scripted telephone call from a diabetes educator or clinical pharmacist to identify and address nonadherence to the new medication or (b) usual care. Hierarchical linear and logistic regression models were used to assess impact on (b) >=2 medication fills within 180 days of prescription,

SECONDARY OUTCOMES:
Composite Control Level of Blood pressure, A1c and/or LDL | 180 days
  In a pragmatic randomized trial, we randomly assigned 2,378 adults with diabetes mellitus who were recently prescribed a new class of medication for elevated glycated hemoglobin (A1c) >= 8%, Blood pressure >= 140/90 mm Hg, or low-density lipoprotein cholesterol >=100 mg/dL, to receive (a) one scripted telephone call from a diabetes educator or clinical pharmacist to identify and address nonadherence to the new medication or (b) usual care. Hierarchical linear and logistic regression models were used to assess impact on (c) clinically significant improvement in a composite measure of A1c, Blood pressure, or low-density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. O'Connor, MD, MPH, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute for Education and Research, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] O'Connor PJ, Schmittdiel JA, Pathak RD, Harris RI, Newton KM, Ohnsorg KA, Heisler M, Sterrett AT, Xu S, Dyer WT, Raebel MA, Thomas A, Schroeder EB, Desai JR, Steiner JF. Randomized trial of telephone outreach to improve medication adherence and metabolic control in adults with diabetes. Diabetes Care. 2014 Dec;37(12):3317-24. doi: 10.2337/dc14-0596. Epub 2014 Oct 14. PMID 25315207